CLINICAL TRIAL: NCT06044792
Title: The Influence of Primary HIV-1 Drug Resistance Mutations on Immune Reconstruction in Patients Treated With Antiretroviral Drugs - an Observational Cohort Study.
Brief Title: The Influence of Primary HIV-1 Drug Resistance Mutations on Immune Reconstruction in PLWH
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: HIV DRM - CD4 reconstruction
Record Dates: First submitted 2023-09-03; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hiv; AIDS; CD4 Deficiency; ART; Treatment Resistant Disorders; Treatment-Sensitive HIV Infection
Keywords: HIV; CD4; DRM; drug resistance; immune reconstruction
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DRM negative: The cohort of patients, who will meet inclusion criteria, with HIV infections and no drug resistance mutations detected.
  Epidemiological (age, sex, origin, sexual preferences) and clinical data (HIV viral load, CD4+ cell count, presence of AIDS-defining diseases, co-infection with HBV and HCV) will be collected at the time of diagnosis.
  Subsequent controls of HIV viral load, level of CD4 and CD4/CD8 ratio will be carried out in accordance with the standard of care for an HIV-infected patient (usually every 6-12 months).
  Interventions: Other: differences in CD4 reconstruction
- DRM positive: The cohort of patients, who will meet inclusion criteria, with HIV infections and detected primary drug resistance mutations.
  Epidemiological (age, sex, origin, sexual preferences) and clinical data (HIV viral load, CD4+ cell count, presence of AIDS-defining diseases, co-infection with HBV and HCV) will be collected at the time of diagnosis.
  Subsequent controls of HIV viral load, level of CD4 and CD4/CD8 ratio will be carried out in accordance with the standard of care for an HIV-infected patient (usually every 6-12 months).
  Interventions: Other: differences in CD4 reconstruction

INTERVENTIONS:
Other: differences in CD4 reconstruction — Differences in the increase in CD4 lymphocyte count and CD4:CD8 ratio between patients with primary drug resistance mutations and those without these mutations.

SUMMARY:
Since the reasons for differential immune reconstitution in HIV-infected patients are still not fully understood, we considered it reasonable to investigate whether the presence of primary HIV drug resistance mutations could be one of the factors of inadequate immune reconstitution.

Evaluation of unfavorable factors of immune reconstitution can help identify patients at risk of persistently low CD4 cell counts and CD4:CD8 ratios and requiring careful monitoring for progression to AIDS.

DETAILED DESCRIPTION:
Untreated HIV infection leads to progressive and permanent impairment of the immune system, and the successive loss of peripheral blood CD4+ T lymphocytes results in progression to AIDS. Effective antiretroviral therapy (ART) can prevent the decline and even cause the restore of the normal level of CD4+ cells.

CD4+ count ≥ 500 cells/µl and CD4:CD8 ratio ≥ 1 are considered normal, while patients with persistently lower CD4+ and CD4:CD8 ratios despite ART treatment are defined as having an inadequate immune response, which may result in an increased risk progression to AIDS, and thus higher mortality rates. Clinical risk factors for impaired CD4+ regeneration have not been fully established, however, older age, male gender, low CD4+ cell count and low CD4:CD8 ratio at diagnosis are associated with a poorer immune response to ART.

As well, HIV drug resistance also plays an important role in the process of immune reconstruction. Despite the very good results of ART, the emergence of drug-resistant mutations in the HIV virus, which may lead to treatment failure, is a cause for concern. The prevalence of HIV-1 drug resistance mutations reported worldwide ranges from 5% to 25%. Primary drug resistance of HIV occurs in people who have not previously been treated with ART. These people start ART treatment with a lower genetic barrier, a higher risk of virological failure and a higher risk of developing resistance to other drugs, which may lead to insufficient immune reconstruction and progression to AIDS.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 confirmed infection
* ART naive patients > 18 years
* virological suppression after 6 months of ART
* available results of HIV genotyping before the start of ART

Exclusion Criteria:

* hematologic neoplasms
* use of chemotherapy, immunosuppressive drugs and other myelotoxic agents
* lack of patient's consent to participate in the study

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will meet the inclusion and not the exclusion criteria will be divided into the 2 groups: with and without DRMs, depending on the results of HIV genotyping. In cohorts subsequent CD4 count and CD4/CD8 ratio will be assessed every 6-12 months in the 4 -year period. Differences in the increase in CD4+ lymphocyte count and CD4:CD8 ratio between patients with primary drug resistance mutations and those without these mutations were taken as the endpoint.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Differences in CD4 recovery regarding the presence of HIV DRM | 4 years
  Differences in the increase in CD4+ lymphocyte (cells/µL) count and CD4:CD8 ratio between patients with primary drug resistance mutations and those without these mutations were taken as the endpoint.

IPD SHARING:
Plan to Share IPD: No
Data will be available on demand to the editors.

REFERENCES:
- [Background] Shenoy N, Ramapuram JT, Shenoy A, Ahmed J, Srikant N. Incidence of Opportunistic Infections among HIV-Positive Adults on Highly Active Antiretroviral Therapy in a Teaching Hospital, India: Prospective Study. J Int Assoc Provid AIDS Care. 2017 May/Jun;16(3):309-311. doi: 10.1177/2325957416686192. Epub 2017 Jan 4. PMID 28050923
- [Background] Gaines H, von Sydow MA, von Stedingk LV, Biberfeld G, Bottiger B, Hansson LO, Lundbergh P, Sonnerborg AB, Wasserman J, Strannegaard OO. Immunological changes in primary HIV-1 infection. AIDS. 1990 Oct;4(10):995-9. doi: 10.1097/00002030-199010000-00008. PMID 2261128
- [Background] Sobrino-Vegas P, Moreno S, Rubio R, Viciana P, Bernardino JI, Blanco JR, Bernal E, Asensi V, Pulido F, del Amo J, Hernando V; Cohorte de la Red de Investigacion en Sida, Spain. Impact of late presentation of HIV infection on short-, mid- and long-term mortality and causes of death in a multicenter national cohort: 2004-2013. J Infect. 2016 May;72(5):587-96. doi: 10.1016/j.jinf.2016.01.017. Epub 2016 Feb 24. PMID 26920789
- [Background] Gazzola L, Tincati C, Bellistri GM, Monforte Ad, Marchetti G. The absence of CD4+ T cell count recovery despite receipt of virologically suppressive highly active antiretroviral therapy: clinical risk, immunological gaps, and therapeutic options. Clin Infect Dis. 2009 Feb 1;48(3):328-37. doi: 10.1086/595851. PMID 19123868
- [Background] Yang X, Su B, Zhang X, Liu Y, Wu H, Zhang T. Incomplete immune reconstitution in HIV/AIDS patients on antiretroviral therapy: Challenges of immunological non-responders. J Leukoc Biol. 2020 Apr;107(4):597-612. doi: 10.1002/JLB.4MR1019-189R. Epub 2020 Jan 22. PMID 31965635
- [Background] Rhee SY, Kassaye SG, Barrow G, Sundaramurthi JC, Jordan MR, Shafer RW. HIV-1 transmitted drug resistance surveillance: shifting trends in study design and prevalence estimates. J Int AIDS Soc. 2020 Sep;23(9):e25611. doi: 10.1002/jia2.25611. PMID 32936523
- [Background] Bokharaei-Salim F, Esghaei M, Khanaliha K, Kalantari S, Marjani A, Fakhim A, Keyvani H. HIV-1 reverse transcriptase and protease mutations for drug-resistance detection among treatment-experienced and naive HIV-infected individuals. PLoS One. 2020 Mar 2;15(3):e0229275. doi: 10.1371/journal.pone.0229275. eCollection 2020. PMID 32119691
- [Background] Grant RM, Hecht FM, Warmerdam M, Liu L, Liegler T, Petropoulos CJ, Hellmann NS, Chesney M, Busch MP, Kahn JO. Time trends in primary HIV-1 drug resistance among recently infected persons. JAMA. 2002 Jul 10;288(2):181-8. doi: 10.1001/jama.288.2.181. PMID 12095382
- [Background] Wensing AM, Calvez V, Ceccherini-Silberstein F, Charpentier C, Gunthard HF, Paredes R, Shafer RW, Richman DD. 2019 update of the drug resistance mutations in HIV-1. Top Antivir Med. 2019 Sep;27(3):111-121. PMID 31634862